CLINICAL TRIAL: NCT01517204
Title: The Comparison of Direct Laryngoscope and Trachway (R) Intubating Stylet in the Insertion of the Double Lumen Endobronchial Tube
Brief Title: The Efficacy of Trachway (R) Intubating Stylet in the Insertion of the Double Lumen Endobronchial Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUH-IRB-990305
Record Dates: First submitted 2011-11-15; First posted 2012-01-25 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2011-05

CONDITIONS: Anesthesia Intubation Complications
Keywords: Trachway(R) intubating stylet; Left sided double lumen endobronchial tube; Efficacy; Intubation complication

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Direct laryngoscope (Experimental): Direct laryngoscope was used to facilitate the intubation of left-sided double lumen endobronchial tube.
  Interventions: Device: Direct laryngoscope (Macintoish laryngoscope)
- Trachway(R) intubating stylet (Experimental): Trachway(R) intubating stylet was used to facilitate left-sided double lumen endobronchial tube intubation.
  Interventions: Device: Trachway(R) intubating stylet

INTERVENTIONS:
Device: Direct laryngoscope (Macintoish laryngoscope) — Direct laryngoscope was used to facilitate the intubation of left-sided DLT.
  Other Names: Macintoish laryngoscope
  Arms: Direct laryngoscope
Device: Trachway(R) intubating stylet — Trachway(R) intubating stylet was used to facilitate the intubation of left-sided DLT.
  Other Names: The Clarus Video System
  Arms: Trachway(R) intubating stylet

SUMMARY:
The purpose of this study is to investigate the effects of Trachway(R) compared with direct laryngoscope in tracheal intubation of double-lumen endobronchial tube.

DETAILED DESCRIPTION:
Intubation with the double-lumen endobronchial tube (DLT) remains a great challenge for anesthesiologists. Although new upper airway devices, such as Trachway (R), a video-assisted intubating stylet, had been developed for facilitating airway management.

The larger size and the complexity of DLT than single-lumen tube (SLT) makes the difficulties for DLT intubation. Therefore, the investigators designed this study to investigate the effects of Trachway(R)compared with direct laryngoscope in DLT intubation.

ELIGIBILITY:
Inclusion Criteria:

1. patients with American Society of Anesthesiologists physical status I-III
2. More than 18 years of age
3. Requiring DLT for thoracic surgery

Exclusion Criteria:

1. risk of regurgitation and pulmonary aspiration
2. history of gastroesophageal reflux, pregnancy
3. scheduled tracheostomy and postoperative prolonged ventilation in ICU
4. patients with limited neck extension (< 35°)
5. a distance between the tip of the patient's mandible and hyoid bone of less than 7 cm
6. a sternomental distance of less than 12.5 cm with the head fully extended
7. mouth can not open

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Main outcome measure is the successful rate of the first intubation | 12 month

SECONDARY OUTCOMES:
The outcome measure is the time needed to insert the DLT | 12 months
The outcome measure is mean blood pressure (MAP) during intubation period | 12 months
  MAP was measured before intubation, and after intubation 1, 3,and 5 min.
The outcome measure is the heart rate (HR) during intubation period | 12 months
  HR was measured and recorded before intubation, and after intubation 1, 3,and 5 min.
The outcome measure is the incidence of hypoxemia. | 12 months
  Hypoxemia was defined as SPO2 less than 90%. Hypoxemia was recorded during the period of intubation.
The outcome measure is the incidence of sore throat. | 12 months
  Sore throat was observed and evaluated after extubation and patient regained consciousness.
The outcome measure is the incidence of hoarseness. | 12 months
  Hoarseness was observed and evaluated after extubation and patient regained consciousness.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Te Hsu, VS, Principal Investigator — Department of anesthesia, Kaoshiung medical university hospital
Locations (1):
- department of anesthesia, Kaohsiung medical university memorial hospital, Kaohsiung City, Kaohsiung, Taiwan